CLINICAL TRIAL: NCT03464877
Title: Prognostic Factors of a Favorable Outcome Following a Supervised Exercise Program for Soldiers With Sub-acute and Chronic Low Back Pain
Brief Title: Prognostic Factors of a Favorable Outcome Following an Exercise Program for Soldiers With Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marc Perron (Other)
Collaborators: Canadian Forces Health Services Centre Ottawa (Other)
Responsible Party: Sponsor-Investigator, Marc Perron, Professor of clinic, Laval University
Organization: Laval University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2012-13-#14
Record Dates: First submitted 2018-02-26; First posted 2018-03-14 (Actual); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Prospective cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): Standardized six-week duration multi-station full-body supervised exercise program. The frequency was 2-3 sessions per week. The duration of each session was 60 minutes.
  Interventions: Other: Multi-station full-body supervised exercise program

INTERVENTIONS:
Other: Multi-station full-body supervised exercise program — The exercise program was 6-week duration, 2-3 visits per week. It was composed of 7 stations, each consisting of numerous exercises of increasing difficulty. The exercises were grouped together as follows: Hip strengthening and control (Station 1); The squat and its variants (Station 2); Elastic bands and the Bodyblade (Station 3); Abdominal planks and their variants (Station 4); Abdominal strengthening (Station 5); Back extensor strengthening (Station 6); and Lifting techniques (Station 7).

SUMMARY:
Low back pain (LBP) encompasses heterogeneous patients unlikely to respond to a unique treatment. Identifying sub-groups of low back pain may help to improve treatment outcomes. Our objective was to identify variables associated with a favorable outcome in soldiers with sub-acute and chronic LBP participating in a multi-station full-body supervised exercise program. The results obtained may permit generation of potential treatment effect modifiers that will eventually have to be validated before being recommended for clinical practice.

DETAILED DESCRIPTION:
All participants took part in the 6-week exercise program, as well as in the two evaluation sessions (pre- and post- exercise program). At the initial evaluation, subjects completed forms and questionnaires on sociodemographics, symptomatology, comorbidities, work restrictions, pain and functional limitations and fear-avoidance beliefs. A physiotherapist measured their lumbar and hip mobility, conducted diagnostic and pain provocation tests and assessed endurance of the trunk muscles. Following the initial evaluation, subjects took part in the 6-week multi-station full-body supervised exercise program (2 to 3 sessions per week). The Oswestry disability questionnaire (ODI) was completed at the initial and at the final evaluations. The change in ODI score following the program was considered the principal measure reflecting favorable or unfavorable outcome.

An improvement of 50% in the initial ODI score was considered the reference standard to determine a favorable outcome. Univariate associations with favorable outcome were tested using chi-square or paired t-tests. Variables that showed between-group (favorable/unfavorable) differences were entered into a logistic regression after determining the sampling adequacy. Finally, continuous variables were dichotomized and the sensitivity, specificity and positive and negative likelihood ratios were determined for the model and for each variable.

ELIGIBILITY:
Inclusion Criteria:

* episode of subacute or chronic LBP with or without radiation to the lower limbs
* minimal score of 17% on the Modified Oswestry Disability Index

Exclusion Criteria:

* previous surgery to the spinal column,
* lumber spine injection in the past two weeks
* signs of upper motor neuron lesions
* serious medical conditions (e.g. tumor, fracture, rheumatoid arthritis, osteoporosis)
* unavailability to participate in the 6-week exercise program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2013-03-19 (Actual); Primary Completion 2015-03-14 (Actual); Study Completion 2015-04-27 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the degree of disability in persons with Low back pain at 6 weeks | Baseline and 6 weeks after the start of the exercises program
  The Modified Oswestry Disability Index is a self-administered questionnaire (10 questions with numerical scale 0-5) whose purpose is to evaluate the severity of the limitations and restrictions suffered by patients with LBP

SECONDARY OUTCOMES:
Height of participants | Baseline
  Tape measure graduated in meter (m)
Weight of participants | Baseline
  On a scale graduated in kilogram (kg)
Body mass index | Baseline
  Weight (kg) divided by the square of the height (m^2) of the participants. Units : Kg/m^2
Fear-Avoidance Beliefs Questionnaire | Baseline
  Self-administered questionnaire that consists of 16 questions (numerical scale 0-6) pertaining to patients' beliefs regarding the effect of their physical activities and work on low back pain
Length of employment in the army | Baseline
  Number of months - (obtained from participants interview)
History of Low Back pain | Baseline
  Dichotomous scale (yes/No) - (obtained from participants interview)
Time since last onset of low back pain | Baseline
  Number of months (obtained from participants interview)
Number of treatments received before initial evaluation in the study | Baseline
  Number of visits (obtained from participants interview)
Referred pain in lower limbs | Baseline
  Dichotomous scale (yes/No) - (obtained from participants interview)
Work restrictions | Baseline
  Nominal scale - three levels (None, less than 6 months, six months or more) - obtained from participants interview)
Sensation of tingling or numbness | Baseline
  Dichotomous scale (yes/No) - (obtained from participants interview)
Use of antidepressant | Baseline
  Dichotomous scale (yes/No) - (obtained from participants interview)
Use of anti-inflammatory drugs | Baseline
  Dichotomous scale (yes/No) - (obtained from participants interview)
Pain in sitting position | Baseline
  Visual analog scale graduated 0-100
Pain in lying position | Baseline
  Visual analog scale graduated 0-100
Pain in standing position | Baseline
  Visual analog scale graduated 0-100
Pain during walking | Baseline
  Visual analog scale graduated 0-100
Pain when coughing or sneezing | Baseline
  Visual analog scale graduated 0-100
Mean pain perceived in the last 48 hours | Baseline
  Visual analog scale graduated 0-10
Worst pain perceived in the last 48 hours | Baseline
  Visual analog scale graduated 0-10
Lumbar and Hip Mobility | Baseline
  Goniometric measurements in degree
Screening or diagnostic tests of lumbar instability | Baseline
  Clinical tests. Dichotomous scale (+/-)
Endurance of the extensor muscles of the trunk | Baseline
  Biering-Sorensen test. Holding time in second
Endurance of the anterior abdominal muscles of the trunk | Baseline
  Abdominal endurance test. Holding time in second
Endurance of the lateral muscles of the trunk | Baseline
  Lateral plank test. Holding time in second

CONTACTS AND LOCATIONS:
Overall Officials: Marc Perron, M.Sc., Principal Investigator — Laval University
Locations (1):
- Laval University, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
The dataset used and/or analysed during the current study is available from the corresponding author on request
Supporting Information: Study Protocol, SAP
Time Frame: upon publication
Access Criteria: on request

REFERENCES:
- [Derived] Perron M, Gendron C, Langevin P, Leblond J, Roos M, Roy JS. Prognostic factors of a favorable outcome following a supervised exercise program for soldiers with sub-acute and chronic low back pain. BMC Musculoskelet Disord. 2018 Apr 2;19(1):95. doi: 10.1186/s12891-018-2022-x. PMID 29606114